CLINICAL TRIAL: NCT05813652
Title: Relative Impacts on Preventative Primary Care--a Longitudinal Evaluation of COVID-19 (Phase 1: A Retrospective Cohort Analysis)
Brief Title: Relative Impacts on Preventative Primary Care--a Longitudinal Evaluation of COVID-19:Phase 1
Acronym: RIPPLE-C
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Michelle Howard, Michelle Howard, PhD, McMaster University
Other Study IDs: WI1-179885
Record Dates: First submitted 2023-04-12; First posted 2023-04-14 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus; Congestive Heart Failure; Chronic Kidney Diseases; Chronic Obstructive Pulmonary Disease; Depression, Anxiety; Osteoarthritis; Dementia
MeSH Terms: conditions — Diabetes Mellitus; Heart Failure; Renal Insufficiency, Chronic; Pulmonary Disease, Chronic Obstructive; Depression; Anxiety Disorders; Osteoarthritis; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- RIPPLE-C cohort: This is a retrospective closed cohort study using a single-arm, pre-post design. Therefore, we will be selecting patients from the CPCSSN database to create our single-arm cohort. Patients included in this cohort will be 18 years of age or older, and will have had at least one contact with their primary care clinic between the dates of March 13, 2018 and March 13, 2020.
  Interventions: Other: Pre-pandemic time period (Jun 22, 2018 to March 12, 2020); Other: Peri-pandemic time period (March 13, 2020 to December 3, 2021)

INTERVENTIONS:
Other: Pre-pandemic time period (Jun 22, 2018 to March 12, 2020) — The primary exposure is the time period of the pandemic (March 13, 2020 to Dec 3, 2021), compared to pre-pandemic (Jun 22, 2018 to pandemic onset March 12, 2020)
Other: Peri-pandemic time period (March 13, 2020 to December 3, 2021) — The primary exposure is the time period of the pandemic (March 13, 2020 to Dec 3, 2021), compared to pre-pandemic (Jun 22, 2018 to pandemic onset March 12, 2020)

SUMMARY:
The goal of this observational study is to describe the impacts of COVID-19 on primary care chronic condition management in Canada within various patient populations. This will be done by analyzing primary care electronic medial record (EMR) data from the Canadian Primary Care Sentinel Surveillance Network (CPCSSN) database, including data on primary care encounters, as well as various markers for chronic conditions.

The research questions to be investigated are:

1a) What are the changes to the management of chronic conditions in primary care since the onset of the COVID-19 pandemic?

1b) How do these changes differ by age, health status, and socioeconomic status?

DETAILED DESCRIPTION:
This is a retrospective closed cohort study, using a single-arm, pre-post design. The objectives of this study are to describe the impacts of COVID-19 on access, comprehensiveness and appropriateness among adult patients with chronic diseases, and to determine whether changes were associated with socio-demographic characteristics and multi-morbidity. This will be done using using electronic medial record (EMR) data made available by the CPCSSN network. CPCSSN is a research network supported by a primary care EMR database, comprising over 1500 physicians, and nearly 2 million patients from across Canada.

We will be examining prevention and management activities for several exemplar chronic conditions that have a validated CPCSSN case definition and substantial prevalence in primary care (e.g. diabetes, heart failure, etc.). CPCSSN data between 2018-2021 will be analyzed for changes in management of various chronic conditions prior to, and through phases of the pandemic. Changes will also be examined among specific sub-groups of adults, including those with multi-morbidity and socio-economic vulnerabilities.

The primary exposure is the onset of the pandemic: March 13, 2020 to December 3, 2021 versus the equal time frame prior. March 13, 2020 was selected as the date when Canadian provincial governments began enforcing various public health and safety measures in response to the World Health Organization formally declaring the circulating SARS-CoV-2 as a pandemic on March 11, 2020.

We will be examining whether there have been changes in overall access, comprehensiveness, continuity and appropriateness of care (including potential decreases in burdensome or unnecessary care) by applying indicators that incorporate chronic condition monitoring (physical measures, lab tests and investigations), prescriptions, referrals and preventive care, to chronic condition patient populations.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older as of 2018
* Records included in the CPCSSN database
* Patient had at least one encounter with their clinic between March 13, 2018 and March 13, 2020

Exclusion Criteria:

* Patients aged 105 or older as of 2018 will be excluded due to possibility of data entry error

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is all patients who were age 18 years and older in 2018. As only year of birth is available, we will use the mid-point of the year for age calculation. We will include patients who have had at least one encounter or form of contact with their primary care clinic between the dates of March 13, 2018 and March 13, 2020. People with a deceased status during the study period will be included up to the point of death.
Sampling Method: Non-Probability Sample
Enrollment: 919928 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Number and types of encounters (access, comprehensiveness) | Beginning of COVID-19 pandemic, March 13, 2020 through December 3, 2021 as compared to an equal time period prior to pandemic start
  Overall number and types of patient encounters; number and types of chronic condition-related encounters for patients with specific chronic conditions (e.g. diabetes, heart failure, etc.). *Note: All outcomes will be measured as applicable to patients' medical conditions and/or age*
Diagnoses addressed in encounters (comprehensiveness, appropriateness) | Beginning of COVID-19 pandemic, March 13, 2020 through December 3, 2021 as compared to an equal time period prior to pandemic start. Where possible, monthly rates will be calculated.
  Overall number of diagnoses addressed per person, per year; number and proportion of encounters for specific chronic conditions addressed at least once a year; number of patients with specific chronic conditions (e.g. diabetes, heart failure, etc.) with condition-related encounters within 6 months, 12 months. *Note: All outcomes will be measured as applicable to patients' medical conditions and/or age.*
Services provided (comprehensiveness) | Beginning of COVID-19 pandemic, March 13, 2020 through December 3, 2021 as compared to an equal time period prior to pandemic start. Where possible, monthly rates will be calculated.
  Number of patients receiving pneumococcal vaccine, influenza vaccine; proportion of patients with specific chronic disease vaccinated for influenza *Note: All outcomes will be measured as applicable to patients' medical conditions and/or age*
Procedures performed (appropriateness) | Beginning of COVID-19 pandemic, March 13, 2020 through December 3, 2021 as compared to an equal time period prior to pandemic start. Where possible, monthly rates will be calculated.
  Proportion of diabetic patients with foot exam in last 12 months *Note: All outcomes will be measured as applicable to patients' medical conditions and/or age*
Physical exams (appropriateness) | Beginning of COVID-19 pandemic, March 13, 2020 through December 3, 2021 as compared to an equal time period prior to pandemic start. Where possible, monthly rates will be calculated.
  Proportion of patients (all patients and those grouped by chronic condition) with blood pressure measured every 6 months, or every 12 months (as appropriate for condition) *Note: All outcomes will be measured as applicable to patients' medical conditions and/or age*
Referrals made to specialists (comprehensiveness) | Beginning of COVID-19 pandemic, March 13, 2020 through December 3, 2021 as compared to an equal time period prior to pandemic start. Where possible, monthly rates will be calculated.
  Overall number of referrals made to specialist providers; proportion of patients with specific chronic condition referred to specific specialties as appropriate based on condition (e.g. endocrinology for diabetic patients, cardiology for heart failure patients, etc.) *Note: All outcomes will be measured as applicable to patients' medical conditions and/or age*
Investigations performed (appropriateness) | Beginning of COVID-19 pandemic, March 13, 2020 through December 3, 2021 as compared to an equal time period prior to pandemic start. Where possible, monthly rates will be calculated.
  Overall number of investigations and laboratory tests; number and frequency of investigations and laboratory tests performed for patients based on presence of chronic conditions (e.g. number of diabetic patients with HbA1C measured every 6 and 12 months) *Note: All outcomes will be measured as applicable to patients' medical conditions and/or age*
Monitoring results (appropriateness) | Beginning of COVID-19 pandemic, March 13, 2020 through December 3, 2021 as compared to an equal time period prior to pandemic start. Where possible, monthly rates will be calculated.
  Proportion of patients with blood pressure below, at, or above target (as appropriate based on age and presence of chronic conditions); number and proportion of patients with systolic blood pressure in the following ranges: <130, 131-140, 141-150, 151-160, >160 *Note: All outcomes will be measured as applicable to patients' medical conditions and/or age*
Medications (appropriateness, comprehensiveness) | Beginning of COVID-19 pandemic, March 13, 2020 through December 3, 2021 as compared to an equal time period prior to pandemic start. Where possible, monthly rates will be calculated.
  Overall number and frequency of medications specific to chronic conditions (e.g. insulin, oral antidiabetics for diabetic patients, angiotensin receptor blockers and/or angiotensin-converting enzyme inhibitors for heart failure patients, etc.); proportion of patients with specific chronic conditions on indicated medications; number of patients who smoke on nicotine replacement therapy *Note: All outcomes will be measured as applicable to patients' medical conditions and/or age*

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Howard, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University Department of Family Medicine, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available to other researchers.

REFERENCES:
- [Derived] Howard M, Freeman K, Hafid S, Vanstone M, Queenan J, Aubrey-Bassler K, Drummond N, Nicholson K, Mangin D. Primary care for depression before and during the COVID-19 pandemic: a retrospective pre-post study. BMJ Open. 2026 Jan 9;16(1):e108681. doi: 10.1136/bmjopen-2025-108681. PMID 41513423
- [Derived] Howard M, Aubrey-Bassler K, Drummond N, Lussier MT, Queenan JA, Vanstone M, Nicholson K, Ramdyal A, Lawson J, Hafid S, Freeman K, Clark R, Mangin D. Effects of the COVID-19 Pandemic on Primary Health Care for Chronic Conditions in Canada: Protocol for a Retrospective Pre-Post Study Using National Practice-Based Research Network Data. JMIR Res Protoc. 2023 Jul 21;12:e49131. doi: 10.2196/49131. PMID 37477967